CLINICAL TRIAL: NCT02985970
Title: Rapid Sequence Induction in Czech Republic: Survey
Brief Title: Rapid Sequence Induction Czech Republic: Survey
Acronym: RSICZ
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Doc.MD.Ph.D, Brno University Hospital
Other Study IDs: RSI 2016CZ
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Rapid Sequence Induction
Keywords: crush induction, RSI
MeSH Terms: conditions — Cumulative Trauma Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ČSARIM - questionnaire: Members of Czech society of anesthesiology, resuscitation and intensive care will obtain the questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — The questionnaire will be send to all members of ČSARIM with the selected 4 controversial clinical scenarios in which the RSI should be used
  Other Names: survey

SUMMARY:
Rapid sequence induction (RSI) is a common part of routine anesthesiology practice.However several steps of RSI are not based on evidence based data (EBM) and are considered controversial. In an electronic evaluation form that will be send to Czech society of anesthesiology, resuscitation and intensive care (ČSARIM) members, the investigators bring 4 clinical scenarios in which RSI should be used. In the questionnaire the participants have to choose RSI or no and they have to describe all the next steps on anesthesia induction process in each single clinical scenario.

DETAILED DESCRIPTION:
Rapid sequence induction (RSI) is a common part of routine anesthesiology practice.However several steps of RSI are not based on evidence based data (EBM) and are considered controversial. In an electronic evaluation form that will be send to Czech society of anesthesiology, resuscitation and intensive care (ČSARIM) members, the investigators bring 4 clinical scenarios in which RSI should be used. In the questionnaire the participants have to choose RSI or no and they have to describe all the next steps on anesthesia induction process in each single clinical scenario.

* 1st. scenario - adult patient with acute abdomen in the OR to be anesthetized
* 2nd. scenario - 4 years old child with acute abdomen in the OR scheduled for an acute surgery
* 3rd. scenario - pregnant women scheduled for an elective caesarean section in the OR
* 4th. scenario - geriatric patient with hiatal hernia scheduled for an elective laparoscopic cholecystectomy.

In each scenario the several steps of the RSI sequence has to be answered:

Is RSI indicated? Y N

Peripheral vein line before induction? Y N

Nasogastric tube before/after induction or without?

Patients position: neutral, head-up, head-down?

Preoxygenation - 3/5minutes, breaths, (CPAP)/Positive end-expiratory pressure (PEEP)?

Sellick manoeuver? Y N

Drugs for induction (order with the number in the row) - propofol, etomidate, ketamine, thiopental, midazolam, suxamethonium, rocuronium, cisatracurium, atracurium, vecuronium

Manual hand-bag ventilation after induction: with limited pressure/contraindicated

Airway: tracheal tube with the cuff/without cuff/laryngeal mask

Comments

ELIGIBILITY:
Inclusion Criteria:

* all members of ČSARIM and www.akutne.cz

Exclusion Criteria:

* not members of ČSARIM and www.akutne.cz

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiologists - members of the ČSARIM and www.akutne.cz
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
RSI practice in Czech Republic - questionnaire | one month
  Evaluation of the clinical practice of the RSI in Czech Republic

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, doc.MD.Ph.D, Study Chair — University Hospital Brno

IPD SHARING:
Plan to Share IPD: Undecided